CLINICAL TRIAL: NCT00005523
Title: Home Based Environmental Adherence Trial
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5050; R18HL058942 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2006-01

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To conduct a randomized trial in asthmatic children to compare the effectiveness of a home-based allergen control program with a customary educational program delivered in offices

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

Two-hundred-forty children, 6 to 17 years of age, were recruited to participate in the study. Following the collection of baseline data, all families in the study received standard environmental control education prior to randomization to the control or experimental group. This education provided parents and children with information about such topics as the child's sensitivity profile, the relationship between exposure to allergens and asthma, and the risks of passive smoking. All families were given information on how to receive environmental control aids and services available by mail at no or reduced costs.

Once families were randomized, those in the control group received no additional intervention. Those in the experimental group received a home-based allergen control intervention delivered by trained environmental counselors. Primary outcomes were changes in asthma-related quality of life and changes in targeted allergen levels in the home. Secondary outcome measures included self-efficacy for environmental allergy control, FEV1, and parent-reported health care utilization.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1998-08; Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peyton Eggleston — Johns Hopkins University

REFERENCES:
- [Background] Eggleston PA. Environmental causes of asthma in inner city children. The National Cooperative Inner City Asthma Study. Clin Rev Allergy Immunol. 2000 Jun;18(3):311-24. doi: 10.1385/CRIAI:18:3:311. No abstract available. PMID 10981263
- [Background] Eggleston PA. Control of environmental allergens as a therapeutic approach. Immunol Allergy Clin North Am. 2003 Aug;23(3):533-47, viii-ix. doi: 10.1016/s0889-8561(03)00003-1. PMID 14524390
- [Background] Matsui EC, Wood RA, Rand C, Kanchanaraksa S, Swartz L, Curtin-Brosnan J, Eggleston PA. Cockroach allergen exposure and sensitization in suburban middle-class children with asthma. J Allergy Clin Immunol. 2003 Jul;112(1):87-92. doi: 10.1067/mai.2003.1588. PMID 12847484
- [Background] Matsui EC, Wood RA, Rand C, Kanchanaraksa S, Swartz L, Eggleston PA. Mouse allergen exposure and mouse skin test sensitivity in suburban, middle-class children with asthma. J Allergy Clin Immunol. 2004 May;113(5):910-5. doi: 10.1016/j.jaci.2004.02.034. PMID 15131574
- [Background] Eggleston PA, Butz A, Rand C, Curtin-Brosnan J, Kanchanaraksa S, Swartz L, Breysse P, Buckley T, Diette G, Merriman B, Krishnan JA. Home environmental intervention in inner-city asthma: a randomized controlled clinical trial. Ann Allergy Asthma Immunol. 2005 Dec;95(6):518-24. doi: 10.1016/S1081-1206(10)61012-5. PMID 16400889